CLINICAL TRIAL: NCT06342193
Title: Effect of Virtual Reality Glasses on Anxiety During Cystoscopy: A Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: virtual reality
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cystoscopy; Virtual Reality; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): This group will use virtual reality glasses during cystoscopy.
  Interventions: Device: virtual reality group
- controlled group (No Intervention): No intervention

INTERVENTIONS:
Device: virtual reality group — This group will use virtual reality glasses as distraction during cystoscopy.
  Arms: intervention group

SUMMARY:
The aim of this study was to investigate the effect of using virtual reality glasses as a distraction method on anxiety in men undergoing cystoscopy under local anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* 18 years of age or older
* Male gender
* undergoing a rigid cystoscopy procedure for the first time
* Application of local anaesthesia

Exclusion Criteria:

* Cognitive or physical disabilities that may prevent the use of virtual reality glasses.
* Premedication before the procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
anxiety | 30 minutes
  State Trait Anxiety Scale-Situational Anxiety Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yucel Can Danisman, Principal Investigator — Usak University Training and Research Hospital
Locations (1):
- Usak Training and Research Hospital, Uşak, Center, Turkey (Türkiye)